CLINICAL TRIAL: NCT07356466
Title: Clinical Efficacy of Pucotenlimab Combined With Lenvatinib and SOX Versus SOX Alone in Patients With HER2-Negative Advanced Gastric or Gastroesophageal Junction Adenocarcinoma: A Single-Center Randomized Controlled Trial
Brief Title: Clinical Efficacy of Pucotenlimab Combined With Lenvatinib and SOX Versus SOX Alone in Patients With HER2-Negative Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: FUGES032
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of Department of Gastric Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES032
Record Dates: First submitted 2025-12-21; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Gastric (Stomach) Cancer
Keywords: Gastric Cancer; HER2-Negative; Objective response rate
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Group (Experimental): Participants receive Study Drug Pucotenlimab Combined with Lenvatinib and SOX .
  Interventions: Drug: Pucotenlimab Combined with Lenvatinib
- Control Group (Other): Oxaliplatin plus S-1 regimen
  Interventions: Drug: Oxaliplatin plus S-1 regimen

INTERVENTIONS:
Drug: Pucotenlimab Combined with Lenvatinib — Pucotenlimab Combined with Lenvatinib
  Arms: Research Group
Drug: Oxaliplatin plus S-1 regimen — Oxaliplatin plus S-1 regimen
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the objective response rate (ORR) of Pembrolizumab combined with Lenvatinib and SOX compared with SOX alone in the treatment of patients with HER2-negative advanced gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
At present, for patients with advanced gastric cancer, palliative chemotherapy or the best supportive care is the main treatment approach, but the therapeutic effect is not satisfactory. The median survival time is around 10-16 months, and the survival rate of patients is very low. How to improve the treatment effect of advanced gastric cancer is an urgent problem to be solved. Currently, several studies on immunotherapy combined with chemotherapy for gastric cancer are underway. From the subgroup analyses of a series of studies ，it can be seen that the expression of PDL1 is increased, which provides a basis for the treatment of advanced tumors with immune checkpoint inhibitors. Studies have shown that the combination of Lenvatinib can reduce angiogenesis in mice, reprogram vascular structure, enhance the infiltration of CD8+ T cells, CD8+ TNFα+ T cells and CD8+ IFNγ+ T cells, and decrease the proportion of MDSCs and macrophages. This provides a basis for the combined use of Lenvatinib and immune checkpoint inhibitors in the treatment of advanced tumors. This study adopts a single-center, prospective research method, aiming to explore the clinical effectiveness and safety of Pucotenlimab combined with Lenvatinib and the SOX regimen in the treatment of patients with HER2-negative advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

**Inclusion Criteria** 1. Age 18-75 years (inclusive). 2. Histologically or cytologically confirmed unresectable, locally advanced or metastatic HER2-negative adenocarcinoma of the stomach or gastro-oesophageal junction (GEJ).

3. No prior systemic chemotherapy, radiotherapy, targeted therapy, or immunotherapy for advanced disease. Subjects who have received prior (neo)adjuvant chemotherapy and/or radiotherapy are eligible provided the last dose was completed ≥ 6 months before randomisation.

4. At least one measurable lesion per RECIST 1.1 (see Appendix 2). 5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1 (see Appendix 4).

6. Estimated life expectancy > 3 months. 7. Adequate major organ function defined as:

1. Haematology (obtained ≤ 14 days without transfusion):

   1. Hb ≥ 80 g/L
   2. WBC ≥ 3 × 10⁹/L
   3. ANC ≥ 1.5 × 10⁹/L
   4. PLT ≥ 100 × 10⁹/L
2. Biochemistry:

   1. Total bilirubin < 1.5 × upper limit of normal (ULN)
   2. ALT and AST < 2.5 × ULN; ALP ≤ 1.5 × ULN
   3. Serum creatinine ≤ 1 × ULN and calculated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula) 8. Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to enrolment and must use highly effective contraception from screening until 8 weeks after the last dose of study drug. Men must be surgically sterile or agree to use effective contraception during the same period.

      9. No participation in any other interventional clinical trial during the pre-treatment or on-treatment phases of this study.

      10. Voluntary written informed consent obtained; willing and able to comply with study procedures and follow-up.

      Exclusion Criteria:

      Exclusion Criteria

      Subjects meeting any of the following conditions will be excluded from enrollment:
      1. Known or suspected hypersensitivity to the investigational drug or any drug of the same class.
      2. Other malignancies within the past 5 years, except adequately treated basal-cell or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix.
      3. Currently receiving treatment in another interventional clinical trial, or any systemic anti-gastric-cancer therapy within 4 weeks prior to the first dose.
      4. Systemic Chinese patent medicines with anti-tumor indications or immunomodulatory agents (e.g., thymosin, interferon, interleukins; local intrapleural use for effusion control is permitted) received within 2 weeks before the first dose.
      5. Prior exposure to: anti-PD-1, anti-PD-L1, anti-PD-L2, or any agent targeting other T-cell co-stimulatory or co-inhibitory pathways (including but not limited to CTLA-4, OX-40, CD137); or prior chemotherapy including S-1.
      6. Live-vaccine administration within 4 weeks before enrollment or planned during the study.

         Note: Inactivated seasonal influenza vaccine by injection is allowed within 4 weeks; intranasal live-attenuated influenza vaccine is prohibited.
      7. Active autoimmune disease requiring systemic therapy (e.g., immunosuppressants, corticosteroids, or disease-modifying agents) within 2 years before the first dose. Replacement therapy (thyroxine, insulin, physiologic glucocorticoids for adrenal or pituitary insufficiency) is not considered systemic therapy.
      8. Prior allogeneic bone-marrow or solid-organ transplantation.
      9. Any condition that could impair drug absorption or inability to swallow oral medication.
      10. Uncontrolled hypertension despite optimal medical management:

          * SBP ≥ 150 mmHg or DBP ≥ 100 mmHg on a single antihypertensive, or requirement of ≥ 2 antihypertensive agents.
      11. Urinalysis showing proteinuria ≥ 2+ and 24-h urinary protein > 1.0 g.
      12. Active gastro-duodenal ulcer, ulcerative colitis, or other gastrointestinal disorders with bleeding risk; un-resected tumors with active hemorrhage; or any other condition judged by the investigator to predispose to GI bleeding or perforation.
      13. Significant bleeding tendency within 3 months before enrollment: overt bleeding > 30 mL, hematemesis, melena, hematochezia; hemoptysis (> 5 mL fresh blood within 4 weeks); or thrombo-embolic event (including stroke/TIA) within 12 months.
      14. Clinically significant cardiovascular disease:

          * Acute MI, unstable/severe angina, or CABG within 6 months before enrollment;
          * NYHA class > II congestive heart failure;
          * Ventricular arrhythmia requiring therapy;
          * QTc ≥ 480 ms on baseline ECG.
      15. Active or uncontrolled severe infection (≥ CTCAE grade 2).
      16. Known HIV infection; clinically significant hepatic disorders:

          * Chronic hepatitis B with active replication (HBV DNA > 1 × 10⁴ copies/mL or > 2000 IU/mL);
          * Hepatitis C with detectable HCV RNA (> 1 × 10³ copies/mL);
          * Other hepatitis or cirrhosis.
      17. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
      18. Any condition that, in the opinion of the investigator, would compromise the subject's safety or interfere with study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 30day
  Objective Response Rate (ORR) is defined as the proportion of patients with confirmed complete response (CR) or partial response (PR) based on standardized, objective criteria (e.g., RECIST 1.1).
Objective Response Rate | 30day
  This study uses the objective response rate (ORR) as the primary efficacy evaluation metric.

SECONDARY OUTCOMES:
Median Overall Survival | according to the OS
  Median Overall Survival (OS) is defined as the time from the date of diagnosis or initiation of treatment to the point at which 50% of patients have died (or reached the study endpoint event), serving as a key indicator for evaluating treatment efficacy and prognosis in chronic diseases such as cancer.
Progression-Free Survival | 36 months
  Progression-Free Survival (PFS) is defined as the time from randomization (or initiation of treatment) to the first documented disease progression (PD) or death from any cause, whichever occurs first
Duration of Response | 30day
  Duration of Response (DOR) is defined as the time from the first documented complete response (CR) or partial response (PR) until disease progression (PD) or death from any cause, whichever occurs first.
Adverse Event | 30 days
  Adverse Event (AE) Incidence Rate is defined as the proportion of participants in a defined analysis set who experience at least one adverse event during a specified observation period after initiation of an intervention (drug, device, or procedure); it quantifies the frequency of intervention-related risk.
Serious Adverse Event | 30 days
  erious Adverse Event (SAE) Incidence Rate is defined as the proportion of participants in a defined analysis set who experience at least one adverse event meeting seriousness criteria during a specified observation period after initiation of an intervention; it quantifies intervention-related risks with potential for major medical consequences or death.
Quality of Life (QoL) assessment | 36 months
  Quality of Life (QoL) assessment is the systematic collection of patients' subjective experience across multiple domains-including physical function, psychological state, social adaptation, and symptom burden-using validated, standardized patient-reported outcome (PRO) instruments; it quantifies the overall impact of disease and its treatment on patients' daily living and serves as a key endpoint in clinical research and therapeutic decision-making.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinrich MC, Jones RL, von Mehren M, Schoffski P, Serrano C, Kang YK, Cassier PA, Mir O, Eskens F, Tap WD, Rutkowski P, Chawla SP, Trent J, Tugnait M, Evans EK, Lauz T, Zhou T, Roche M, Wolf BB, Bauer S, George S. Avapritinib in advanced PDGFRA D842V-mutant gastrointestinal stromal tumour (NAVIGATOR): a multicentre, open-label, phase 1 trial. Lancet Oncol. 2020 Jul;21(7):935-946. doi: 10.1016/S1470-2045(20)30269-2. PMID 32615108
- [Background] Tang X, Yang J, Shi A, Xiong Y, Wen M, Luo Z, Tian H, Zheng K, Liu Y, Shu C, Ma N, Wang R, Zhao J. CD155 Cooperates with PD-1/PD-L1 to Promote Proliferation of Esophageal Squamous Cancer Cells via PI3K/Akt and MAPK Signaling Pathways. Cancers (Basel). 2022 Nov 15;14(22):5610. doi: 10.3390/cancers14225610. PMID 36428703
- [Background] Lai X, Gupta SK, Schmitz U, Marquardt S, Knoll S, Spitschak A, Wolkenhauer O, Putzer BM, Vera J. MiR-205-5p and miR-342-3p cooperate in the repression of the E2F1 transcription factor in the context of anticancer chemotherapy resistance. Theranostics. 2018 Jan 1;8(4):1106-1120. doi: 10.7150/thno.19904. eCollection 2018. PMID 29464002
- [Background] Furtado J. Decentralising HIV treatment in lower- and middle-income countries. Sao Paulo Med J. 2014 Dec;132(6):383. doi: 10.1590/1516-3180.20141326t2. PMID 25351762
- [Background] Wang W, Kirsch T. Annexin V/beta5 integrin interactions regulate apoptosis of growth plate chondrocytes. J Biol Chem. 2006 Oct 13;281(41):30848-56. doi: 10.1074/jbc.M605937200. Epub 2006 Aug 16. PMID 16914549
- [Background] Goser S, Ottl R, Brodner A, Dengler TJ, Torzewski J, Egashira K, Rose NR, Katus HA, Kaya Z. Critical role for monocyte chemoattractant protein-1 and macrophage inflammatory protein-1alpha in induction of experimental autoimmune myocarditis and effective anti-monocyte chemoattractant protein-1 gene therapy. Circulation. 2005 Nov 29;112(22):3400-7. doi: 10.1161/CIRCULATIONAHA.105.572396. PMID 16316965
- [Background] Paulus BC, Adelman SL, Jamula LL, McCusker JK. Leveraging excited-state coherence for synthetic control of ultrafast dynamics. Nature. 2020 Jun;582(7811):214-218. doi: 10.1038/s41586-020-2353-2. Epub 2020 Jun 11. PMID 32528090
- [Background] Hasson A, Jiang W, Benabdallah N, Lu P, Longtine MS, Beattie BJ, Summer L, Zhang H, Wahl RL, Abou DS, Thorek DLJ. Radiochemical Quality Control Methods for Radium-223 and Thorium-227 Radiotherapies. Cancer Biother Radiopharm. 2023 Feb;38(1):15-25. doi: 10.1089/cbr.2022.0023. Epub 2022 Sep 23. PMID 36149725
- [Background] Walczak-Sztulpa J, Wawrocka A, Doornbos C, van Beek R, Sowinska-Seidler A, Jamsheer A, Bukowska-Olech E, Latos-Bielenska A, Grenda R, Bongers EMHF, Schmidts M, Obersztyn E, Krawczynski MR, Oud MM. Identical IFT140 Variants Cause Variable Skeletal Ciliopathy Phenotypes-Challenges for the Accurate Diagnosis. Front Genet. 2022 Jul 7;13:931822. doi: 10.3389/fgene.2022.931822. eCollection 2022. PMID 35873489
- [Background] Zhu YZ, Zhong JX, Dong LL. Menstrual and Reproductive Characteristics of Patients with Primary Sjogren's Syndrome: A 7-year Single-center Retrospective Study. Curr Med Sci. 2023 Feb;43(1):139-145. doi: 10.1007/s11596-022-2675-4. Epub 2022 Dec 21. PMID 36542325
- [Background] Monga J, Adrianto I, Rogers C, Gadgeel S, Chitale D, Alumkal JJ, Beltran H, Zoubeidi A, Ghosh J. Tribbles 2 pseudokinase confers enzalutamide resistance in prostate cancer by promoting lineage plasticity. J Biol Chem. 2022 Feb;298(2):101556. doi: 10.1016/j.jbc.2021.101556. Epub 2021 Dec 30. PMID 34973338
- [Background] Bhowmick T, Liu C, Imp B, Sharma R, Boruchoff SE. Ceftaroline as salvage therapy for complicated MRSA bacteremia: case series and analysis. Infection. 2019 Aug;47(4):629-635. doi: 10.1007/s15010-019-01304-7. Epub 2019 Apr 6. PMID 30955166
- [Background] Wang SM, Han C, Lee SJ, Jun TY, Patkar AA, Masand PS, Pae CU. Investigational dopamine antagonists for the treatment of schizophrenia. Expert Opin Investig Drugs. 2017 Jun;26(6):687-698. doi: 10.1080/13543784.2017.1323870. Epub 2017 May 12. PMID 28443355
- [Background] Zhang MZ, Yao B, Wang S, Fan X, Wu G, Yang H, Yin H, Yang S, Harris RC. Intrarenal dopamine deficiency leads to hypertension and decreased longevity in mice. J Clin Invest. 2011 Jul;121(7):2845-54. doi: 10.1172/JCI57324. Epub 2011 Jun 23. PMID 21701066
- [Background] Craig A, Kool J, Nilles E. The Pacific experience: supporting small island countries and territories to meet their 2012 International Health Regulations (2005) commitments. Western Pac Surveill Response J. 2013 Jul 3;4(3):14-8. doi: 10.5365/WPSAR.2012.3.4.007. eCollection 2013 Jul-Sep. PMID 24319608
- [Background] Luo H, Li S, Zhao M, Sheng B, Zhu H, Zhu X. Prognostic value of progesterone receptor expression in ovarian cancer: a meta-analysis. Oncotarget. 2017 May 30;8(22):36845-36856. doi: 10.18632/oncotarget.15982. PMID 28415663
- [Background] Ostergaard KH, Bertelsen MF, Brondum ET, Aalkjaer C, Hasenkam JM, Smerup M, Wang T, Nyengaard JR, Baandrup U. Pressure profile and morphology of the arteries along the giraffe limb. J Comp Physiol B. 2011 Jul;181(5):691-8. doi: 10.1007/s00360-010-0545-z. Epub 2011 Jan 5. PMID 21207038
- [Background] Puza CJ, Warren WS, Mosca PJ. Correction to: The changing landscape of dermatology practice: melanoma and pump-probe laser microscopy. Lasers Med Sci. 2017 Dec;32(9):2173. doi: 10.1007/s10103-017-2339-y. PMID 28980190
- [Background] Liu Y, Zhou K, Guo S, Wang Y, Ji X, Yuan Q, Su L, Guo X, Gu X, Xing J. NGS-based accurate and efficient detection of circulating cell-free mitochondrial DNA in cancer patients. Mol Ther Nucleic Acids. 2021 Jan 1;23:657-666. doi: 10.1016/j.omtn.2020.12.017. eCollection 2021 Mar 5. PMID 33575112
- [Background] Almeida GJ, Khoja SS, Zelle BA. Effect of prehabilitation in older adults undergoing total joint replacement: An Overview of Systematic Reviews. Curr Geriatr Rep. 2020 Dec;9(4):280-287. doi: 10.1007/s13670-020-00342-6. Epub 2020 Nov 24. PMID 33344110
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338